CLINICAL TRIAL: NCT03759418
Title: Left Atrial Appendage Ligation Using the Atriclip Device; Single Center Study of Device Safety and Efficacy
Brief Title: Left Atrial Appendage Ligation Using the Atriclip Device
Status: Completed | Type: Observational
Sponsor: St. Helena Hospital Coon Joint Replacement Institute (Other)
Collaborators: AtriCure, Inc. (Industry); Adventist Heart and Vascular Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 005
Record Dates: First submitted 2018-09-10; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-09

CONDITIONS: Left Atrial Appendage Ligation
Keywords: Left Atrial Appendage Ligation; Atriclip; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: exclusion of the left atrial appendage — A trans esophageal echocardiogram will be performed to assess the Atriclip device in the closure of the left atrial appendage in patients that had surgery at least 12 months ago.

SUMMARY:
The purpose of the study is to collect data regarding ligation of the left atrial appendage at least 12 months after surgery for patients that had exclusion of the left atrial appendage as a primary minimally invasive procedure or in conjunction with other open cardiac or minimally invasive cardiac procedures.

DETAILED DESCRIPTION:
The purpose of this study is to collect data regarding ligation of the left atrial appendage at least 12 months after surgery for patients that had exclusion of the left atrial appendage as a primary minimally invasive procedure or in conjunction with other open cardiac or minimally invasive cardiac procedures. The patient will undergo a transesophageal echocardiogram (TEE) to collect the following data: Left Ventricular Ejection Fraction; Left Atrial diameter size; confirmation of Left Atrial Appendage exclusion defined by the absence of left atrial to LAA (left atrial appendage) communication measured in millimeters and absence of LAA pocket measured in millimeters; presence of thrombus in left atrium.

ELIGIBILITY:
Inclusion Criteria:

* All adult patient who had a heart procedure where an Atriclip device was deployed as the primary or secondary procedure between 3/2013-12/20/2016
* Patient is willing to undergo a trans esophageal echocardiogram, or if unable a CT angiogram
* If female, must be of non-childbearing potential or have a negative pregnancy test within 7 days prior to the procedure
* Patient is willing to sign an IRB approved Informed Consent

Exclusion Criteria:

* Patient did not have an Atriclip device as part of the surgical procedure between 3/2013 and 12/2016.
* Patient is unwilling or unable to undergo trans esophageal echocardiogram with general anesthesia or a CT angiogram

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who had an Atriclip placed to exclude the left atrial appendage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
12 month follow up with complete exclusion of the Left Atrial Appendage | 365 days to complete
  The complete exclusion is defined by the lack of fluid communication between the left atrium and left atrial appendage at </= 12 months

SECONDARY OUTCOMES:
Any signs of thrombus in the left atrium | 365 days to compete
  Any signs of thrombus in the left atrium
Occurrence of Cerebrovascular accident/transient Ischemic Attack | 365 days to complete
  Occurrence of Cerebrovascular accident/transient ischemic attack postoperative ,/= 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gansevoort Dunnington, MD, Principal Investigator — St. Helena Hospital Adventist Heart Institute

IPD SHARING:
Plan to Share IPD: No